CLINICAL TRIAL: NCT00662324
Title: Development of a Clinical Trial Specific Question Prompt List
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-042; NIH/NCI R03 CA130598-01
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Lung Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1: Trial experienced cancer patients and their primary caregivers.
  Interventions: Behavioral: focus groups
- 2: Trial naive cancer patients and their caregivers.
  Interventions: Behavioral: focus groups
- 3: Health care professionals who are involved in running Phase I, II or III clinical trials.
  Interventions: Behavioral: focus groups

INTERVENTIONS:
Behavioral: focus groups — Focus group with MSKCC patients with lung, breast and prostate cancer who have taken part in clinical trials and other caregivers. This focus group will be audio recorded.
  During the focus group, you will discuss a Question Prompt List that will be handed out to you. You will be asked about what you think of it and if you think it would have been useful to the patient you care for in his/her experience in a clinical trial.
  The focus group to last from 60 to 90 minutes.
  Groups: 1
Behavioral: focus groups — Focus group with MSKCC patients with lung, breast and prostate cancer who have not taken part in clinical trials and other caregivers. This focus group will be audio recorded.
  During the focus group, you will discuss a Question Prompt List that will be handed out to you. You will be asked about what you think of it and if you think it would be useful if the patient you care for were ever to take part in a clinical trial sometime in the future.
  We expect the focus group to last from 60 to 90 minutes.
  Groups: 2
Behavioral: focus groups — MSKCC clinicians who work with lung, breast and prostate cancer patients. This focus group will be audio recorded.
  During the focus group, you will discuss a Question Prompt List that will be handed out to you. You will be asked about what you think of it and if you think it would be useful to your patients who take part in clinical trials.
  Expect the focus group to last from 60 to 90 minutes.
  Groups: 3

SUMMARY:
The purpose of this study is to develop a Question Prompt List (QPL) about clinical trials for cancer patients and find out what cancer patients and their caregivers think of the QPL. A QPL is a list of questions patients might want to ask their doctors during their appointments.

We will conduct three focus groups to talk about using QPL's as a new way to recruit patients like you to clinical trials. The three groups will be made of patients who have and have not participated in clinical trials, their caregivers and doctors. This study is also being done to learn about how the QPL affects the question asking behavior of patients during their appointments with doctors at Memorial SloanKettering Cancer Center (MSKCC).

ELIGIBILITY:
Inclusion Criteria:

* Population Segment 1 who have participated in a clinical trial
* Diagnosis and treatment at MSKCC of lung, prostate or breast cancer
* Completion of a Phase I, II, or III clinical trial at MSKCC
* Ability to provide informed consent

Patient caregiver eligibility requirements will be:

* Nomination by patient as the primary caregiver
* Ability to provide informed consent

Population Segment 2 who have not participated in a clinical trial:

* Diagnosis and treatment at MSKCC of lung, prostate or breast cancer or the primary patient caregiver
* Ability to provide informed consent

Patient caregiver eligibility requirements will be:

* Nomination by patient as the primary caregiver
* Ability to provide informed consent

Population Segment 3 who are health care professionals:

* A current health care professional at MSKCC
* Current involvement in recruiting patients with lung, prostate or breast cancer to Phase I,II, or III clinical trials at MSKCC
* Ability to provide informed consent

Exclusion Criteria:

Potential subjects will be considered ineligible for either/both phases of this study if they are:

* Fewer than 18 years of age
* Cognitively or physically impaired, rendering them incapable of providing informed consent to participate in the study
* Population Segment 2 participants will be excluded if they have ever participated in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: treatment at MSKCC of lung, prostate or breast cancer A current health care professional at MSKCC current involvement in recruiting patients with lung, prostate or breast cancer to Phase I,II, or III clinical trials at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2008-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To develop a targeted Question Prompt List for Clinical Trials and evaluate its acceptability to cancer patients considering clinical trial participation. | conclusion of study

SECONDARY OUTCOMES:
To explore the utility of the Question Prompt List for Clinical Trials in oncology consultations containing a discussion of a Phase I, II or III clinical trial. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Bylund, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org